CLINICAL TRIAL: NCT01482793
Title: A Controlled Trial of Vertebroplasty for Acute Painful Osteoporotic Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optimus Clinical Research (Other)
Collaborators: C. R. Bard (Industry)
Responsible Party: Principal Investigator, Paul Bird, Principal Investigator, Optimus Clinical Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WGT4P; VAPOUR (Other: Other)
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Vertebral Compression Fractures; Osteoporotic Vertebral Compression Fractures; Acute Vertebral Fractures
MeSH Terms: interventions — Vertebroplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AVAMAX (Active Comparator): Avamax vertebroplasty kits provided by Care Fusion
  Interventions: Procedure: Vertebroplasty
- Simulated injection procedure (No Intervention): Patient will be unaware as to whether the control procedure or vertebroplasty had been performed since full sterile preparation, sedation and simulated injection procedure will be used.

INTERVENTIONS:
Procedure: Vertebroplasty — AVAmax radiopaque bone cement is injected into the vertebral body using a 13 G or 11 G vertebroplasty needle.
  Arms: AVAMAX

SUMMARY:
The objective of this study is to gather data regarding the efficacy, safety and cost-effectiveness of percutaneous vertebroplasty in the acute fracture group with fractures less than 6 weeks old. The AVAMAX vertebroplasty kits (Care Fusion) will be used for all vertebroplasties.

The primary effectiveness analysis will be based on the number of patients whose numeric rating pain score drops from above 7 out of 10 at baseline to below 4 out of 10 at two weeks post-intervention. Our hypothesis is that the vertebroplasty group will have a significantly larger proportion of patients achieving pain reduction than the control group. A secondary analysis will compare the change in mean pain scores and specific activity related pain scores between the two groups at 3 days, 14 days and at 1, 3 and 6 months. Another secondary effectiveness analysis will include the mean change in the back-pain specific limitation in function as quantified by the Roland Scale at these same data collection time points.

DETAILED DESCRIPTION:
The study will be a two arm randomised, blind placebo controlled trial of vertebroplasty for acute (< 6 weeks) osteoporotic vertebral compression fractures. Patients with substantial pain or immobility despite medical therapy will be recruited to the study, randomised to study treatments and followed for 6 months. The primary effectiveness variable is back-pain as recorded on a numerical verbal rating scale at two weeks post-procedure. Secondary effectiveness variable will be the Roland Morris back pain specific disability score.

In parallel with the trial an economic analysis will be conducted.

Study participants will be recruited from patients who are referred for vertebroplasty evaluations from five clinical sites of the Sydney metropolitan area. The sites will be St George Private Hospital, Kareena Private Hospital, St George Public Hospital, Sutherland Hospital and Liverpool Hospital. These sites have the advantage of having robust, established vertebroplasty programs and high levels of technical operator experience with vertebroplasty in acute fractures. Potential patients are patients identified with a recent vertebral fracture that requires assessment for a vertebroplasty. The referring physician will request an MRI and spinal radiograph as part of routine assessment and standard clinical care. Potential involvement in the study will be discussed at this point between patient and referring physician. Patients will be given a consent form to read and consider. The research team will then contact potential subjects and ask them a series of questions to determine eligibility. The investigator and the research coordinator will then describe the study to eligible patients and informed consent will be obtained prior to conducting baseline evaluations and randomization.

Treatment Intervention (Vertebroplasty Procedure):

5.1.1 The procedure is performed under strict aseptic conditions. All personnel wear surgical masks and caps in addition to gowns and gloves for operators, to minimize the risk of infection. 1G ceftriaxone will be administered at the commencement of the procedure unless the patient is allergic. In case of allergy then antibiotics are not mandatory.

5.1.2 The patient is placed prone on the angiographic table and oxygen mask applied. Conscious sedation will be induced by IV administration of fentanyl and midazolam.

5.1.3 Continuously monitor heart rate and pulse oximetry throughout the procedure.

5.1.4 Standard fluoroscopy with a dedicated DSA interventional fluoroscope will be used for localization of the vertebral body to be treated (Levels T4-L5) and needle placement within the vertebral body.

5.1.5 A 25g needle will be used to raise a wheal of 1% lignocaine subcutaneously. A small skin nick will be made with a scalpel blade. A 25g needle will be placed into the skin at the site of the wheal and advanced under fluoroscopic guidance to the periosteum over the pedicle. This periosteum will be infiltrated with 6-7 cc of 1% lignocaine. (Injections will be made at each fracture level, i.e., 2 separate injections will be performed for patients with 2 fracture levels.) 5.1.6 A small incision is made on the skin in the vicinity of the pedicle, and the access needle is positioned for a transpedicular approach.

5.1.7 13G or 11G vertebroplasty needles will be placed using trans-pedicular or para-pedicular approach into the anterior one third of the vertebral body. Whether a unilateral or bilateral approach is used is up to the discretion of the radiologist doing the procedure, but a bi-pedicular approach is recommended for the T12 vertebral body and all of the lumbar vertebral bodies (due to their increased size). An effort should be made to fill both the fractured fragment of the vertebral body and the more normal trabecular component in order to stop ongoing fracture and volume loss.

5.1.8 Prepare the AVAMAX™ injecting system in the approved manner as per system instruction. Wait for 5 minutes after mixing cement before cement injection to allow for optimal viscosity prior to commencing injection. Product accountability forms will be completed which include batch numbers.

5.1.9 Cement injection should be performed using continuous fluoroscopic screening in the lateral projection. Cement injection should continue until adequate vertebral body filling is obtained. This ideally means cement filling from the superior to inferior vertebral body end-plate in at least the anterior three quarters of the vertebral body in lateral projection. In frontal projection, the cement should reach at least from middle of the pedicle to middle of the contra-lateral pedicle in a distribution considered adequate (by the radiologist) to stabilize the acute fracture. Upon completion of injection, the cannula is removed and haemostasis at the puncture site is achieved by gentle pressure. If adequate fill was not obtained, place another needle in the contra lateral pedicle and treat in the same fashion.

5.1.10 Patient should be left in prone position for 3 minutes following cement injection to allow for cement to harden.

5.1.11 Contingency plans should an outpatient have a sudden life threatening event occur in the radiology suite and require immediate medical or surgical attention: patient will be examined and appropriate life support measures instituted. In case of suspected spinal cord compromise, immediate CT scanning and surgical consultation will be made. In the case of hemodynamic compromise from idiosyncratic reaction, life support will be instituted.

5.2 Control Intervention: 5.2.1 The procedure is performed under strict aseptic conditions. All personnel wear surgical masks and caps in addition to gowns and gloves for operators, to minimize the risk of infection and to simulate a true vertebroplasty. Prophylactic antibiotics may be administered by the treating physician according to their usual practice, but are not mandated by the study protocol.

5.22 The patient is placed prone on the angiographic table and oxygen mask applied. Conscious sedation will be induced by IV administration of fentanyl, morphine or pethidine and midazolam.

5.2.3 Continuously monitor heart rate and pulse oximetry throughout the procedure.

5.2.4 Standard fluoroscopy will be used for localization of the vertebral body to be treated (Levels T4-L5) and needle placement within the vertebral body.

5.2.5 A 25g needle will be used to raise a wheal of 1% lignocaine subcutaneously. A skin incision measuring approximately 5mm will be made. The 25G needle will then be reintroduced and 2 cc of 1% lignocaine injected into the subcutaneous tissues.. (These sham injections will be made at each fracture level, i.e., 2 separate injections will be performed for patients with 2 fracture levels.) 5.2.6 Verbal clues will be given, including but not limited to comments that needle placement and/or cement injection is progressing appropriately. Manual palpation of the area over the fracture will be done to simulate needle placement.

5.2.8 The procedure will be terminated.(Note: The patient will be unaware as to whether the control procedure or vertebroplasty had been performed since full sterile preparation, sedation and simulated injection procedure will be used.

5.2.9 Contingency plans should an outpatient have a sudden life threatening or limb threatening event occur in the radiology suite and require immediate medical or surgical attention: patient will be examined and appropriate life support measures instituted. In case of suspected spinal cord compromise, immediate CT scanning and surgical consultation will be made. In the case of hemodynamic compromise from idiosyncratic reaction life support will be instituted.

5.3 Post Operative Care: 5.3.1 Following the procedure, all patients should be observed in the supine position for at least one hour.

5.3.2 Patients may gradually sit up and/or stand over the next hour, as tolerated, under direct nursing or physician supervision.

5.3.3 Outpatients may be discharged to the care of an adult after 2 hours. 5.3.4 Non-narcotic pain medication may be taken as needed, but patients are encouraged to limit use of narcotics so efficacy can be determined.

5.3.5 One hour after the procedure, patients are evaluated for pain, or complications of the procedure. Vital signs will also be recorded.

5.3.6 If determined to be necessary by the physician, an outpatient may be admitted and monitored overnight in the hospital. The reason for keeping the patient overnight will be documented on the post treatment assessment form and the serious adverse event form.

5.3.7 Evaluation of any potential complication will be conducted immediately so that appropriate treatment can be instituted.

5.3.8 Dressings applied to the injection/incision site may be removed the following day.

5.3.9 Skin incisions should be kept clean and dry. Patients are to notify physician of any redness or discharge.

5.3.10 Inpatients will continue to be managed by attending physician in usual fashion.

5.4 Patient Evaluations & Follow Up Examinations We will administer the following measures of pain and pain-related disability questionnaires: numeric and visual pain-rating scale, the Roland-Morris Low Back Pain and Disability Questionnaire, Osteoporosis Quality of Life Questionnaire (QUALEFFO), SF-36 and EQ-5D to all subjects in this trial. We will also ask patients about their use of medications, other health care resources, medical history, co-morbidities and demographics. A timed up and go test, which is a reliable measure of function in older people, will be completed during patient clinic visits at baseline, day 14 and month 6 .

After obtaining informed consent during the baseline consultation, patients will be asked about demographic information and the patient questionnaires will be administered in a face-to-face interview. The two week and six month interviews will also be asked in person by research staff during patient visits. The other interviews (Days 3, day 7, weeks 4 and month 3) will be conducted by telephone for all participants at all sites. An exception to this will be inpatients that remain in hospital at day 3 who may be interviewed at bedside*.

ELIGIBILITY:
Inclusion Criteria/Exclusion Criteria:

* Patient is greater than 60 years of age.
* Patient has pain which is not adequately controlled by oral analgesia or which has required hospitalisation and prevents early mobilisation
* Patient has pain from one or two compression fractures of the vertebrae in the areas T4 to L5 confirmed with a sagittal STIR (short tau inversion recovery) and sagittal T1 weighted MRI scan of the spine. Patients with three or more recent fractures are excluded.
* Clinical history verifies that patient's fracture occurred in the previous 6 weeks.
* Patient does not have a known coagulopathy. If on warfarin, the INR should be less than 2.5 within the last three days.
* Patient has no contraindications for conscious sedation.
* Patient reports pain during ambulation or movement from the compression fracture(s) of at least seven (7) out of ten (10) on a numerical pain scale.
* Patient has access to a telephone.
* Patient speaks English well enough to answer all health questions via telephone.
* Patient has a confirmed diagnosis of osteoporosis via a BMD within 6 months of baseline or a QCT at baseline.
* Patient does not have a history of debilitating chronic back pain which requires regular analgesia.
* Patients with chronic back pain who regularly use medication containing any narcotic for a period greater than 6 weeks, that is prior to the acute fracture.
* Patient does not have significant retropulsed fragment or spinal canal compromise of greater than 20% by retropulsed fragment.
* Patient has no mental incapacity or dementia that makes him/her unable to give informed consent.
* Patient has no history of vertebral osteomyelitis.
* Patient has vertebral body collapse not greater than 60% relative to closest intact vertebra.
* Patient has no pedicle fractures.
* Patient has no active local or systemic infection.
* Patient has not had surgery (within the last 60 days).
* Patient has no concomitant hip fracture.
* Patient has no malignant tumour deposit (multiple myeloma), tumour mass, or tumour extension into the epidural space at the level of the fracture to be treated on MRI.
* Patient does not have severely immunocompromised health status (including any patient who is HIV positive, currently on chemotherapy, taking high doses of long term corticosteroids - defined as a dose of prednisone exceeding 10mg for greater than 3 months in the last 12 months, has a hematologic malignancy, or a transplant recipient.)
* Patient able to attend face to face visits.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Patient rated pain intensity | two weeks

SECONDARY OUTCOMES:
Functional Disability | two weeks
  Functional Disability (Roland Morris disability score) will be measured at 3 days, 7 days, 1 month, 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: William Clark, Principal Investigator — St George Private Hospital
Locations (1):
- Optimus Clinical Research, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Clark W, Bird P, Gonski P, Diamond TH, Smerdely P, McNeil HP, Schlaphoff G, Bryant C, Barnes E, Gebski V. Safety and efficacy of vertebroplasty for acute painful osteoporotic fractures (VAPOUR): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 1;388(10052):1408-1416. doi: 10.1016/S0140-6736(16)31341-1. Epub 2016 Aug 17. PMID 27544377
- [Derived] Clark W, Bird P, Diamond T, Gonski P. Vertebroplasty for acute painful osteoporotic fractures (VAPOUR): study protocol for a randomized controlled trial. Trials. 2015 Apr 12;16:159. doi: 10.1186/s13063-015-0671-8. PMID 25873274